CLINICAL TRIAL: NCT04013711
Title: Quantitative Thermal Imaging to Evaluate Skin Toxicity From Radiation Treatment
Brief Title: Thermal Imaging to Evaluate Skin Toxicity From Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. William Tran, Clinical scientist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 187-2018
Record Dates: First submitted 2018-10-15; First posted 2019-07-10 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2022-02

CONDITIONS: Radiotherapy Side Effect; Radiodermatitis
MeSH Terms: conditions — Radiation Injuries; Radiodermatitis | interventions — Thermography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thermal Imaging (Experimental): Patients will undergo non-invasive, thermal imaging of their whole breast or head and neck cancer site, during the course of the radiotherapy treatment, at weekly time intervals.
  Interventions: Diagnostic Test: Thermography

INTERVENTIONS:
Diagnostic Test: Thermography — Thermograms will be acquired of both treated and non-treated cancer site for comparison.

SUMMARY:
A significant proportion of patients treated with whole-breast or head and neck radiotherapy will experience skin toxicity, i.e. skin dermatitis, which may lead to erythema, dry desquamation and wet desquamation. It is hypothesized that quantitative thermal imaging can be used to measure radiation-induced skin toxicity.

DETAILED DESCRIPTION:
The aim of this study is to use quantitative thermal imaging to evaluate skin toxicity in patients treated with whole-breast or head and neck radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-confirmed diagnosis of breast cancer (Stage 0-III) or head and neck cancer (all subtypes; stage I - IV) according to American Joint Committee on Cancer staging criteria.
2. Subjects must give appropriate written informed consent prior to participation in the study
3. Subjects must be able and willing to comply and understand the instructions associated with the imaging procedure.
4. Both men and women are eligible for participation
5. Subjects must be at least 18 years of age
6. Subjects must be receiving radiotherapy:

   1. adjuvant radiotherapy to the whole breast or chest wall, or;
   2. in the case of head and neck treatment, either as definitive treatment or adjuvantly.
7. definitive radiotherapy of the head and neck

Exclusion Criteria:

1. Subjects with any pre-existing dermatologic abnormalities (open sores, keloids, psoriasis) involving the treated breast or head and neck.
2. Patients with very hairy skin surface (this does not permit measuring the heat output)
3. Subjects with a current or past medical history of connective tissue disease.
4. Subjects who are pregnant or lactating (which usually preclude them from radiotherapy)
5. Subjects, who, in the opinion of the investigator or clinical research coordinator, may not otherwise be appropriate for inclusion into the study, such as significant anxiety, history of musculoskeletal disease which may predispose them to discomfort during the imaging/scanning period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Temperature changes in skin during radiotherapy. | 1 year
  To measure the temperature changes in skin during each week of radiation therapy and correlate to radiotherapy treatment time.

SECONDARY OUTCOMES:
Measure patient-reported toxicity using a validated self-assessment tool (Dermatology Quality of Life Questionnaire) | 1 year
  Measure patient-reported symptoms using a validated questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: William T Tran, PhD, Principal Investigator — Clinician Scientist
Locations (1):
- Sunnybrook Hospital, Toronto, Ontario, Canada